CLINICAL TRIAL: NCT04564664
Title: High-flow Oxygen Therapy During Exercise in Idiopathic Pulmonary Fibrosis: a Crossover Clinical Trial
Brief Title: High-flow Oxygen Therapy During Exercise in Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2017/7397/I
Record Dates: First submitted 2020-09-14; First posted 2020-09-25 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2020-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: exertional desaturation; high-flow nasal cannula
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-flow nasal cannula oxygen therapy (Other)
  Interventions: Drug: Oxygen
- Standard oxygen therapy (Other)
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — High-flow nasal cannula oxygen therapy vs. standard oxygen therapy

SUMMARY:
Objectives:

1. To evaluate endurance time during cardiopulmonary exercise test (CPET) performance comparing standard oxygen therapy to high-flow nasal cannula (HFNC) oxygen therapy in subjects with idiopathic pulmonary fibrosis (IPF) with exertional desaturation.
2. To assess oxygenation level (peripheral and muscular) as well as dyspnea and fatigue during exercise in IPF subjects with exertional desaturation using oxygen supplementation with HFNC compared with standard oxygen supplementation.

Method: multicenter crossover clinical trial. Patients with IPF presenting oxygen desaturation during the six-minute walking test (6MWT) (SpO2 mean ≤ 85%) will be included consecutively . Each subject evaluated will perform initially an incremental CPET to evaluate the patient's maximum exercise capacity. Supplemental oxygen will be applied to maintain SpO2 >85% with a Venturi mask. Maximum exercise capacity and the appropriate final oxygen inspiratory fraction (FiO2) needed for the following tests will be determined.

Posteriorly each patient will perform two constant load CPET (at 75% of the maximum workload achieved with the incremental CPET); one with standard oxygen therapy and the other one with HFNC oxygen therapy. Endurance time, dyspnea and leg fatigue and oxygen saturation (peripheral and muscular) will be recorded.

Evaluation measures: Endurance time, dyspnea and leg fatigue (Borg scale), and oxygen saturation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with IPF diagnosis according to the 2018 international consensus guidelines
* Mean SpO2 ≤ 85% during the 6MWT performed under room air conditions

Exclusion Criteria:

* Fibrotic interstitial lung diseases other than IPF
* Chronic obstructive pulmonary disease (COPD)
* Inability to perform a complete CPET due to osteo-articular or cognitive limitations
* End-stage lung disease
* Severe pulmonary hypertension

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Endurance time | through study completion, an average of 1 week
  Endurance time (s) during the constant load CPET performance with standard oxygen therapy compared to HFNC oxygen therapy

SECONDARY OUTCOMES:
Dyspnea and fatigue | through study completion, an average of 1 week
  Dyspnea and fatigue (Borg scale) at the end of the constant load CPET with standard oxygen therapy compared to HFNC oxygen therapy
Oxygen saturation | through study completion, an average of 1 week
  Peripheral oxygen saturation (SpO2) during the constant load CPET with standard oxygen therapy compared to HFNC oxygen therapy
Muscle oxygen saturation (StO2) | through study completion, an average of 1 week
  Muscle oxygen saturation (StO2) during the constant load CPET with standard oxygen therapy compared to HFNC oxygen therapy

CONTACTS AND LOCATIONS:
Overall Officials: Eva Balcells Vilarnau, Principal Investigator — Hospital del Mar; Diego Agustín Rodriguez Chiariadia, Study Director — Hospital del Mar
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No